CLINICAL TRIAL: NCT02208141
Title: Determinants of Adipose Tissue Development and Obesity in Children and Adolescents
Brief Title: Leipzig Adipose Tissue Childhood Cohort
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Antje Koerner, Prof. Dr. med., Prof. Dr. med., University of Leipzig
Other Study IDs: IFB ADI K7-10
Record Dates: First submitted 2014-06-12; First posted 2014-08-04 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Childhood Obesity; Insulin Resistance
Keywords: children; obesity; adipose tissue dysfunction; inflammation; macrophage infiltration; insulin resistance; dyslipidemia
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Obesity; Inflammation; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * adipose tissue sample
  * mRNA from adipose tissue samples, adipocytes, stromal vascular fraction
  * protein from whole adipose tissue samples
  * blood samples for DNA analysis, serum samples
  * urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lean and obese children and adolescents: study cohort may be stratified for lean (definded as BMI <1.28 SDS) and overweight/obese (definded as BMI>= 1.28 SDS) children for posthoc analyses no intervention

SUMMARY:
In this study the investigators hypothesize that pathological alterations in adipose tissue biology already occur during the development and progression of obesity in children and adolescents. The investigators aim to identify and characterize mechanisms and molecular targets that affect the development of adipose tissue and ensuing obesity in childhood and adolescence.

DETAILED DESCRIPTION:
The investigators aim to identify how adipose tissue dysfunction in childhood contributes to the development of obesity and related comorbidities and to characterize factors that play a role in the development of adipose dysfunction in children. The investigators will employ a translational approach which is based on the characterization of adipose tissue biology in samples of children to determine alterations leading to adipose tissue dysfunction. These include assessment of the composition (including BAT), remodeling, function, metabolism and inflammation of adipose tissue as well as the adipokine profile. For the assessment of clinical relevance, these experimental data will then be correlated with the clinical phenotype. Finally, we aim to identify factors responsible for early adipose tissue dysfunction and characterize them for their clinical and functional relevance.

ELIGIBILITY:
Inclusion Criteria:

* body weight: 3000 g - 180 kg
* suitable surgical procedure
* signed informed consent by the guardians and the study participant, if older 12 years

Exclusion Criteria:

* severe chronic and inflammatory diseases
* acute or chronic infections
* oncological diseases
* clotting disorders
* complications during surgical procedure
* drug treatment
* nil by mouth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: children and adolescents undergoing surgery at the University Hospital Leipzig
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-10; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue dysfunction | 10 years
  Adipose tissue dysfunction is assessed by evaluation of adipocyte size and number (hypertrophy vs. hyperplasia), adipocyte proliferation and differentiation, (lipid) cellular metabolism, inflammation, gene expression, fibrosis, and others; the association of AT dysfunction with clincial phenotype will be assessed

SECONDARY OUTCOMES:
Presence of brown adipose tissue (BAT) | 10 years
  Adipose tissue samples will be evaluated for the presence of BAT on histological and molecular level and association with clinical phenotype will be investigated
Inflammation of adipose tissue | 10 years
  Inflammation will be assessed by evaluating macrophage infiltration on histological and molecular expression level. Also, association with clinical phenotype will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Körner, Prof. Dr., Principal Investigator — University of Leipzig
Locations (1):
- Center for Pediatric Research Leipzig (CPL), Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Kempf E, Landgraf K, Vogel T, Spielau U, Stein R, Raschpichler M, Kratzsch J, Kiess W, Stanik J, Korner A. Associations of GHR, IGF-1 and IGFBP-3 expression in adipose tissue cells with obesity-related alterations in corresponding circulating levels and adipose tissue function in children. Adipocyte. 2022 Dec;11(1):630-642. doi: 10.1080/21623945.2022.2148886. PMID 36384443
- [Derived] Loffler D, Landgraf K, Rockstroh D, Schwartze JT, Dunzendorfer H, Kiess W, Korner A. METRNL decreases during adipogenesis and inhibits adipocyte differentiation leading to adipocyte hypertrophy in humans. Int J Obes (Lond). 2017 Jan;41(1):112-119. doi: 10.1038/ijo.2016.180. Epub 2016 Oct 17. PMID 27748745
- See also: Link to Prof. Dr. med. Antje Körner's research group: "childhood obesity" — http://kik.uniklinikum-leipzig.de/kikcms.site,postext,childhood-obesity-antje-koerner,a_id,1062.html
- See also: Link to University Children's Hospital Leipzig — http://kik.uniklinikum-leipzig.de/